CLINICAL TRIAL: NCT05417802
Title: Surveying Patient's Interest in Robotic Rehabilitation Device
Status: Active, not recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Amit Kandel, MD, MBA, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00004756
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke with acute stroke: Inclusion criteria
  * Episode of single stroke within the past twelve weeks
  * Individuals' age over 18 years old.
  Exclusion criteria
  * Pregnant women , neurological disorders other than stroke (i.e. Parkinson's), non-ischemic stroke
  * Individuals with severe cognitive impairments (demonstrating difficulty to understand, read, and answer the questions in writing)
  * Individuals with difficulties to listen the instruction and video of the robotic device

SUMMARY:
This is a survey study to understand the stroke survivor's interest in robotic training. Investigators will use a questionnaire and show a video of robotic therapy to ask questions on their interest.

DETAILED DESCRIPTION:
The purpose of this research is to investigate the interest of individuals with recent stroke in robotic therapy. Investigators will introduce a novel robotic platform to train ADLs of stroke patients. Investigators will examine the usability of this device as a home trainer for training rotational hand manipulation tasks such as opening a pickle jar, turning a key, missing a pot with a ladle, etc. The device will especially target stroke patients with ischemic stroke to enhance the performance of ADL. Also, investigators will examine the frequency and dosage of the current occupational therapy, followed by the satisfaction of the current therapy. Participant's participation will contribute to the development of a new therapy method using a robotic device for home-based training.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stroke
* Adults with no cognitive difficulties

Exclusion Criteria:

* Adults with pregnancy,
* Adults with other neurological disorders than stroke
* Adults with hemorrhagic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Current Therapy question - 1 | through study completion, an average of 1 year
  How many hours are you receiving occupational therapy for each session?
Current Therapy question - 2 | through study completion, an average of 1 year
  How frequent are you receiving therapy (ex.: 2/week: two times per week)?
Current Therapy question - 3 | through study completion, an average of 1 year
  When did you start your therapy (how many days after stroke)?
Current Therapy question - 4 | through study completion, an average of 1 year
  What kind of therapy are you receiving now?
Current Therapy question - 5 | through study completion, an average of 1 year
  Do you think that the therapy you are receiving is helpful to restore your arm function and help you participate in activities during daily living (example: drinking, feeding, moving objects)?
Current Therapy question - 6 | through study completion, an average of 1 year
  Do you think that you are receiving enough occupational therapy to help you participate in activities during daily living (example: drinking, feeding, moving objects)?
Interest in Robotic Rehabilitation question - 1 | through study completion, an average of 1 year
  Do you think that this device can be helpful to improve your arm function from stroke?
Interest in Robotic Rehabilitation question - 2 | through study completion, an average of 1 year
  Do you think that you will use the device for home training when it is provided?
Interest in Robotic Rehabilitation question - 3 | through study completion, an average of 1 year
  Do you think that the device is helpful to help you participate in activities during daily living (example: drinking, feeding, moving objects)?
Interest in Robotic Rehabilitation question - 4 | through study completion, an average of 1 year
  If you have the device at home, how long would you like to exercise with the device?
Interest in Robotic Rehabilitation question - 5 | through study completion, an average of 1 year
  If you have the device at home, how frequent would like to use this device?
Interest in Robotic Rehabilitation question - 6 | through study completion, an average of 1 year
  Do you think that the training can be more effective by adding virtual reality?
Interest in Robotic Rehabilitation question - 7 | through study completion, an average of 1 year
  If the device can apply therapeutic force, which type of force do you prefer for home-training?

CONTACTS AND LOCATIONS:
Overall Officials: Jiyeon Kang, Principal Investigator — University at Buffalo
Locations (1):
- Buffalo General Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be shared upon request to PI.
Time Frame: After the study is completed
Access Criteria: The personnel who is requesting the data needs to explain how the data will be used in their research.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05417802/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05417802/ICF_001.pdf